CLINICAL TRIAL: NCT01097356
Title: The Effect of Probiotics on the Clearance of the Human Papillomavirus and on Cytological Lesions Caused by the Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Veronique Verhoeven, professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2414VV
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: HPV-related Cytological Abnormalities on PAP Smear (LSIL)
MeSH Terms: conditions — Squamous Intraepithelial Lesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- common care (No Intervention): HPV+ patients with LSIL on their PAP smear, waiting for 6 months to receive a new PAP smear
- probiotic drinkers (Experimental): HPV+, LSIL patients who will drink the study drink for 6 months
  Interventions: Dietary Supplement: probiotic drinkers

INTERVENTIONS:
Dietary Supplement: probiotic drinkers — HPV+, LSIL patients in this arm will drink the probiotic study drink for a period of 6 months
  Arms: probiotic drinkers

SUMMARY:
Aim: In this project proposition the investigators would like to examine the effect of immune modulation by probiotics on the clearance of HPV-infections.

This study provides a model for viral infection but also for cancer precursors. This would be an excellent model (and the only possible short-term model) to examine an effect on cancer precursors. Cancer precursors (cytological abnormalities such as L-SIL) are a scientifically accepted surrogate endpoint for cervical cancer, for example in HPV-vaccine studies.

Research question: Does daily intake of probiotics lead to a better immune-response in HPV-infected women, i.e. does it facilitate clearance of the virus and/or regression of cytological lesions?

ELIGIBILITY:
Inclusion Criteria:

* women with a new LSIL diagnosis an HPV positivity on PAP smear

Exclusion Criteria:

* women over 65
* immunocompromised patients (because of disease or drugs)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
1.proportion of HPV positives in both arms | 6months
2. proportion of regression of LSIL lesion in both arms | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: veronique verhoeven, MD, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Veronique Verhoeven, Wilrijk, Belgium